CLINICAL TRIAL: NCT05736783
Title: Comparative Effects of Plyometric and Strength Training of Quadriceps and Hamstrings on Sprint and Agility Performance in Football Players
Brief Title: Plyometric and Strength Training of Quadriceps and Hamstrings in Football Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0427
Record Dates: First submitted 2023-01-22; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Football Players
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- plyometric exercises (Experimental): performing plyometric exercises for 6 weeks
  Interventions: Other: plyometric exercises
- strenghtening of quadriceps and hamstring (Experimental): performing strengthening of quadriceps and hamstring for 6 weeks
  Interventions: Other: strenghtening of quadriceps and hamstring

INTERVENTIONS:
Other: plyometric exercises — 1. st week Wall touches 3x30 s Split squat jumps 2x40 Lateral cone jumps 2x30 Cone hops with 180 turn 4conesx10
  2. nd week Wall touches 4x30 s Split squat jumps 2x40 Lateral cone jumps 2x30 Cone hops with 180 turn 4 cones x 30
  3. rd week Wall touches 5x30 s Split squat jumps 2x60 Lateral cone jumps 2x50 Cone hops with 180 turn 4 cones x 30
  4. th week Wall touches 5x30 s Split squat jumps 2x60 Lateral cone jumps 2x50 Cone hops with 180 turn 4 cones x 30 Drop jump 45.72 cm 45.72 cm (20)
  5. th week Wall touches 5x30 s Split squat jumps 2x60 Lateral cone jumps 2x50 Cone hops with 180 turn 4 cones x 30 Drop jump 45.72 cm 45.72 cm (30)
  6. th week Wall touches 6x30 s Split squat jumps 2x70 Lateral cone jumps 2x60 Cone hops with 180 turn 4 cones x 40 Drop jump 45.72 cm (40)
  Arms: plyometric exercises
Other: strenghtening of quadriceps and hamstring — 1st to 3rd week l 4th to 6th week Squat 2x12 3x8 l 3x10 4x6 Knee extension 3x12 3x8 l 2x10 2x6 Nordic hamstring 3x3 3x3 l 3x4 3x4
  Arms: strenghtening of quadriceps and hamstring

SUMMARY:
Football is a trendy sport in the world. A typical footballer runs more than 10 kilometers in an average game of 90 minutes. FIFA regulates the sport of football and the world cup is conducted every 4 years. Plyometric exercise training uses speed and different forced movements to build muscle power. Plyometrics training improves physical performance and the ability to do different activities. Strengthening exercises are designed to increase the strength of specific groups of muscles. Strengthening exercises overload the muscle until the point of muscle fatigue. By conducting the study, it will help us to make a better understanding that whether plyometrics or strength training is more effective so that we can cooperate it into the regular exercise of the football player so that their sports performance can be enhanced.

DETAILED DESCRIPTION:
It will be a randomized clinical trial. It will be conducted at the Pakistan sports board and coaching center, Lahore. A sample of 40 athletes will be taken using convenient sampling. Athletes will be randomly allocated into two groups. Group A was given plyometrics and group B was given strengthening exercises. Athletes will be assessed using a 20m sprint test and an Illinois agility test before the initiation of the exercise regimen. Athletes will perform plyometrics 5 days a week and strength training twice a week for 6 weeks. Athletes will be reassessed after 6 weeks. Statistical analysis will be used to determine their effects with the help of the software SPSS 25.

ELIGIBILITY:
Inclusion Criteria:

* the age group of 15-30 years.
* Participants that are practicing five times a week
* Participants having experience of at least 1 year

Exclusion Criteria:

* Athletes with any musculoskeletal injuries;
* Athletes with any systemic illness;
* Novice football players
* Elite/ International players

Ages: 15 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2022-01-08 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
20 meter sprint test | 6 weeks
  20 meter sprint test: a popular test used to determine how fast athlete can run
Illinois Agility Test | 6 weeks
  Illinois Agility Test is a commonly used test of agility in sports

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Asrar Yousaf, Masters, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No